CLINICAL TRIAL: NCT02252939
Title: Factors Associated With Radiographic Pathophysiology for Trapeziometacarpal Arthrosis in Patients Not Seeking Care for This Condition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Neal Chung-Jen Chen, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013P000827
Record Dates: First submitted 2014-08-12; First posted 2014-09-30 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Trapeziometacarpal Arthrosis
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with Trapeziometacarpal (TMC) Arthrosis (Experimental): Patients presenting to the Orthopaedic Hand Service not seeking care for TMC Arthrosis
  Interventions: Radiation: X-Ray

INTERVENTIONS:
Radiation: X-Ray — X-ray as part of standard care

SUMMARY:
The investigators are doing this research study to discover factors, such as job, hobbies, or race that are associated with arthrosis at the base of your thumb on X-rays. Thumb arthrosis is one of the most common kinds of arthritis. About 116 people will take part in this research study at Massachusetts General Hospital (MGH).

ELIGIBILITY:
Inclusion Criteria:

* 55 years and older
* Not seeking care for TMC arthrosis from hand surgeon at the time of visit
* english fluency and literacy

Exclusion Criteria:

-

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-09; Primary Completion 2016-07 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Chen, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Allegrante JP, Marks R. Self-efficacy in management of osteoarthritis. Rheum Dis Clin North Am. 2003 Nov;29(4):747-68, vi-vii. doi: 10.1016/s0889-857x(03)00060-7. PMID 14603581
- [Background] Bijsterbosch J, Visser W, Kroon HM, Stamm T, Meulenbelt I, Huizinga TW, Kloppenburg M. Thumb base involvement in symptomatic hand osteoarthritis is associated with more pain and functional disability. Ann Rheum Dis. 2010 Mar;69(3):585-7. doi: 10.1136/ard.2009.104562. Epub 2010 Feb 2. PMID 20124359
- [Background] Buckelew SP, Parker JC. Coping with arthritis pain. A review of the literature. Arthritis Care Res. 1989 Dec;2(4):136-45. doi: 10.1002/anr.1790020408. PMID 2487718
- [Background] Dahaghin S, Bierma-Zeinstra SM, Ginai AZ, Pols HA, Hazes JM, Koes BW. Prevalence and pattern of radiographic hand osteoarthritis and association with pain and disability (the Rotterdam study). Ann Rheum Dis. 2005 May;64(5):682-7. doi: 10.1136/ard.2004.023564. Epub 2004 Sep 16. PMID 15374852
- [Background] Das De S, Vranceanu AM, Ring DC. Contribution of kinesophobia and catastrophic thinking to upper-extremity-specific disability. J Bone Joint Surg Am. 2013 Jan 2;95(1):76-81. doi: 10.2106/JBJS.L.00064. PMID 23283376
- [Background] DeGood DE, Tait RC. Assessment of pain beliefs and pain coping. In: Turk DC, Melzack R (Eds.) Handbook of pain assessment, 2nd ed. New York, Guilford Press, 2001: 320-45.
- [Background] Dolce JJ, Crocker MF, Moletteire C, Doleys DM. Exercise quotas, anticipatory concern and self-efficacy expectancies in chronic pain: a preliminary report. Pain. 1986 Mar;24(3):365-372. doi: 10.1016/0304-3959(86)90122-3. PMID 3960576
- [Background] Haara MM, Heliovaara M, Kroger H, Arokoski JP, Manninen P, Karkkainen A, Knekt P, Impivaara O, Aromaa A. Osteoarthritis in the carpometacarpal joint of the thumb. Prevalence and associations with disability and mortality. J Bone Joint Surg Am. 2004 Jul;86(7):1452-7. doi: 10.2106/00004623-200407000-00013. PMID 15252092
- [Background] Hoffman BM, Papas RK, Chatkoff DK, Kerns RD. Meta-analysis of psychological interventions for chronic low back pain. Health Psychol. 2007 Jan;26(1):1-9. doi: 10.1037/0278-6133.26.1.1. PMID 17209691
- [Background] Jensen MP, Turner JA, Romano JM, Karoly P. Coping with chronic pain: a critical review of the literature. Pain. 1991 Dec;47(3):249-283. doi: 10.1016/0304-3959(91)90216-K. PMID 1784498
- [Background] Lorig K, Chastain RL, Ung E, Shoor S, Holman HR. Development and evaluation of a scale to measure perceived self-efficacy in people with arthritis. Arthritis Rheum. 1989 Jan;32(1):37-44. doi: 10.1002/anr.1780320107. PMID 2912463
- [Background] Lozano-Calderon SA, Souer JS, Jupiter JB, Ring D. Psychological differences between patients that elect operative or nonoperative treatment for trapeziometacarpal joint arthrosis. Hand (N Y). 2008 Sep;3(3):271-5. doi: 10.1007/s11552-008-9098-y. Epub 2008 Mar 29. PMID 18780109
- [Background] Marshall M, van der Windt D, Nicholls E, Myers H, Dziedzic K. Radiographic thumb osteoarthritis: frequency, patterns and associations with pain and clinical assessment findings in a community-dwelling population. Rheumatology (Oxford). 2011 Apr;50(4):735-9. doi: 10.1093/rheumatology/keq371. Epub 2010 Dec 6. PMID 21134961
- [Background] Ring D, Guss D, Malhotra L, Jupiter JB. Idiopathic arm pain. J Bone Joint Surg Am. 2004 Jul;86(7):1387-91. doi: 10.2106/00004623-200407000-00005. PMID 15252084
- [Background] Sodha S, Ring D, Zurakowski D, Jupiter JB. Prevalence of osteoarthrosis of the trapeziometacarpal joint. J Bone Joint Surg Am. 2005 Dec;87(12):2614-2618. doi: 10.2106/JBJS.E.00104. PMID 16322609
- [Background] Vranceanu AM, Barsky A, Ring D. Psychosocial aspects of disabling musculoskeletal pain. J Bone Joint Surg Am. 2009 Aug;91(8):2014-8. doi: 10.2106/JBJS.H.01512. PMID 19651964
- [Background] Wolf JM, Delaronde S. Current trends in nonoperative and operative treatment of trapeziometacarpal osteoarthritis: a survey of US hand surgeons. J Hand Surg Am. 2012 Jan;37(1):77-82. doi: 10.1016/j.jhsa.2011.10.010. Epub 2011 Nov 25. PMID 22119601

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With Trapeziometacarpal (TMC) Arthrosis
Started | 62
Completed | 59
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Trapeziometacarpal (TMC) Arthrosis
Number analyzed (Participants) | 59
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 67 [61 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 56
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 59

OUTCOME MEASURES:

1. Primary Outcome: Factors Associated With Eaton Classification of Trapeziometacarpal Arthrosis: Age
Description: Radiographs were scored using the Eaton score range.The Eaton score ranges from 1-4 where 1 is the least severe and 4 is the most severe for arthritis. Patients without TMC Arthritis would have a score of 0. Patients' age measured in years.
Time Frame: Baseline at Day 1
Population: Patients presenting to the Orthopaedic Hand Service not seeking care for TMC Arthrosis
  X-Ray: X-ray as part of standard care
Measure: Median (Inter-Quartile Range); unit: Years
Groups:
- Patients With Trapeziometacarpal Arthrosis Eaton Stage I: Patients presenting to the Orthopaedic Hand Service not seeking care for TMC Arthrosis, Eaton Stage I
  X-Ray: X-ray as part of standard care
- Patients With Trapeziometacarpal Arthrosis Eaton Stage II: Patients presenting to the Orthopaedic Hand Service not seeking care for TMC Arthrosis, Eaton Stage II
  X-Ray: X-ray as part of standard care
- Patients With Trapeziometacarpal Arthrosis Eaton Stage III-IV: Patients presenting to the Orthopaedic Hand Service not seeking care for TMC Arthrosis, Eaton Stage III-IV
  X-Ray: X-ray as part of standard care
Arm/Group | Patients With Trapeziometacarpal Arthrosis Eaton Stage I | Patients With Trapeziometacarpal Arthrosis Eaton Stage II | Patients With Trapeziometacarpal Arthrosis Eaton Stage III-IV
Number analyzed (Participants) | 5 | 36 | 18
Years | 61 [56 to 66] | 66 [62 to 70] | 75 [66 to 82]

2. Secondary Outcome: Factors Associated With Thumb Pain: Hyperextension of Metacarpophalangeal Joint
Description: Thumb pain measured on a scale of 0-10 and dichotomized by having thumb pain (yes/no), hyperextension dichotomized (yes/no)
Time Frame: Day 1, baseline
Population: All patients with TMC Arthrosis analyzed for hyperextension of MCP joint.
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Thumb Pain; Patients Without Thumb Pain: Patients presenting to the Orthopaedic Hand Service not seeking care for TMC Arthrosis with thumb pain
  X-Ray: X-ray as part of standard care
Arm/Group | Patients With Thumb Pain | Patients Without Thumb Pain
Number analyzed (Participants) | 11 | 48
Participants | 10 | 26

3. Secondary Outcome: QuickDASH (Disability of the Arm, Shoulder, and Hand)
Time Frame: Day 1, baseline
Population: Data were not collected
Arm/Group | Patients With Trapeziometacarpal (TMC) Arthrosis
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Patients With Trapeziometacarpal (TMC) Arthrosis
Serious Adverse Events (participants affected / at risk) | 0/59
Other Adverse Events (participants affected / at risk) | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes